CLINICAL TRIAL: NCT02318966
Title: A Comparison of Glycosade® and Uncooked Cornstarch (UCCS) for the Dietary Management of Hepatic Glycogen Storage Diseases (GSD)
Brief Title: Glycosade v UCCS in the Dietary Management of Hepatic GSD
Acronym: Glyde
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: University College London Hospitals (Other); University of Florida (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Medical Center Groningen (Other); Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MCTW-GLY-03/14-18
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycosade (Active Comparator): Participants will be randomised to receive the medical food Glycosade as a starch load with a maximum dose of 100g. Glycosade to be taken as one dose.
  Interventions: Dietary Supplement: Medical Food - Glycosade
- Uncooked corn starch (Placebo Comparator): Participants will be randomised to receive uncooked corn starch as a starch load with a maximum dose of 100g. Uncooked corn starch to be taken as one dose.
  Interventions: Dietary Supplement: Medical Food - Glycosade

INTERVENTIONS:
Dietary Supplement: Medical Food - Glycosade — double blind randomised crossover of 2 starches - glycosade and UCCS

SUMMARY:
To compare efficacy of Glycosade® with uncooked corn starch (UCCS for the dietary management of hepatic glycogen storage diseases (GSD).

DETAILED DESCRIPTION:
'Glyde' is a prospective, randomised, double-blind, crossover trial to compare the effects of two different starches used in the dietary management of GSD.

The study will recruit 64 patients from six centres in the UK, USA, France and The Netherlands. The planned duration per participant is 2 years.

Participants will be randomised into two equally sized groups:

Arm A- Glycosade intake given first, followed by UCCS 1-6 weeks later Arm B- UCCS intake given first, followed by Glycosade 1-6 weeks later.

The objective of this trial is to establish whether Glycosade® improves outcomes for patients with GSD compared to UCCS therapy by comparing the duration of normal blood sugars, lactate and ketone levels of patients with hepatic GSD (Types I, III, VI and IX) post equivalent intakes of UCCS and Glycosade®.

The first part consists of two (blinded) 12 hour starch load tests administered randomly within a maximum 6 week period. Participants will be randomised to receive either UCCS or Glycosade® for the initial intervention period crossing over to the other product for the second intervention period (part 1).

The second part (unblinded) is a 24 month open follow up whereby participant's will continue on the product considered most suitable by the clinician and patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by either genetic mutation analysis or enzymology study (this includes patients with only a single mutation but who also have supportive enzymology consistent with the condition). For those whom mutation analysis is not completed this will be assessed during the study.
* Aged 2 years or older (5 years or older in the USA)
* Established on full intake of uncooked corn starch therapy for at least 6 months

Exclusion Criteria:

* Women who are pregnant or breastfeeding at the start of the study or planning to become pregnant during the study will be excluded.
* children less than 2 years of age

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
To assess if Glycosade® will result in improved blood glucose, lactate and ketone levels in a larger group of patients with GSD I, III, VI & IX as measured by duration of normal blood glucose levels or prevention of ketosis | 24 hours

SECONDARY OUTCOMES:
1. The insulin area under the curve during dietary management with UCCS compared to dietary management with Glycosade®. | 24 hours
2. The area under the curve in lactate, BOHB, during dietary management with UCCS compared to dietary management with Glycosade®. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mundy, MRCP MRCPCH, Principal Investigator — Guys and St Thomas NHS Foundation Trust
Locations (6):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States
- Hôpital Antoine Béclère, Clamart, France
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- United Kingdom (3):
  - National Hospital for Neurology and Neurosurgery, London, Greater London
  - Evelina Children's Hospital, London
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No